CLINICAL TRIAL: NCT05687838
Title: The Effect of Two Different Types of Music Applied During Chemotherapy on Anxiety, Nausea and Satisfaction Levels
Brief Title: The Effect of Music Applied During Chemotherapy on Anxiety, Nausea and Satisfaction Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Öznur ERBAY DALLI, Asst. Prof., Uludag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022-13/18
Record Dates: First submitted 2022-12-29; First posted 2023-01-18 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Anxiety; Chemotherapy Effect; Satisfaction, Patient; Cancer; Nursing Caries
Keywords: Music; Chemotherapy; Nursing; Anxiety
MeSH Terms: conditions — Anxiety Disorders; Patient Satisfaction; Neoplasms | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Relaxing Music Group (Experimental): The patients in this group will listen to specially composed "MusiCure®" compositions, which contain melodies with soft rhythm (60-80 bpm), including harp, cello, strings, and nature sounds (such as rain, bird, forest sound). The patients scheduled to receive chemotherapy for the first time, will be allowed to listen to music for at least one hour during chemotherapy with over-ear headphones (Sennheiser HD280) and an MP3 player. Anxiety and satisfaction levels of the patients will be recorded before and after the music application.
  Interventions: Other: Music
- Turkish Makam Music Group (Active Comparator): The patients in this group will listen to the "Rast Makam", which was created as a result of research conducted by the Turkish Music Research and Promotion Group (TÜMATA) and provides individuals with comfort and inner peace. The patients scheduled to receive chemotherapy for the first time, will be allowed to listen to music for at least one hour during chemotherapy with over-ear headphones (Sennheiser HD280) and an MP3 player. Anxiety and satisfaction levels of the patients will be recorded before and after the music application.
  Interventions: Other: Music
- Control Group (No Intervention): The patients in this group will not receive any musical interventions and will receive standard treatment and care during chemotherapy.

INTERVENTIONS:
Other: Music — Music medicine
  Arms: Relaxing Music Group; Turkish Makam Music Group

SUMMARY:
Chemotherapy is a treatment that uses natural or synthetic chemicals and biological agents to kill rapidly proliferating cells. As chemotherapeutic drugs prevent the growth and proliferation of cancer cells, they also inhibit the growth of normal cells such as intestinal and oral mucosal epithelium, bone marrow cells, and hair follicle cells. During chemotherapy treatment, which is widely used in the treatment of cancer cases and considered one of the most effective methods of cancer treatment, individuals; may experience side effects such as nausea-vomiting, loss of appetite, mouth ulcers, pain, fatigue, anxiety, depression, sleep problems, and changes in their skin and nails.

There are several factors that can trigger anxiety in cancer patients: fear of cancer and its treatment-related side effects, fear of relapse after treatment, uncertainty, concerns about changing roles and relationships, and fear of death. Treatment methods are available for a variety of side effects and negative effects experienced by cancer patients. These methods include pharmacological and nonpharmacological approaches. For example, benzodiazepines are frequently used to treat anxiety in cancer patients. If benzodiazepines are not adequate, low-dose antipsychotics can be used. However, benzodiazepines and their derivatives may reduce respiratory function, induce sedation, and cause confusion.

Music is an example of non-pharmacological cognitive-behavioral treatment that is used to control negative symptoms in many fields. The use of music for healing is easy, has no side effects, and is beneficial for physical, psychological, emotional, and spiritual well-being. Anxiety and fear can be reduced by therapeutic music, which increases endorphin secretion and positive emotions. Treatment of serious illnesses such as cancer requires a holistic approach that includes psychological, social, and spiritual support in addition to pharmacological treatment. Therefore, the purpose of this study is to examine how different types of music affect cancer patients' anxiety and satisfaction during chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old,
* Receiving chemotherapy for the first time.

Exclusion Criteria:

* Hearing or vision problems,
* Have a lower education level than secondary school (The STAI is appropriate for those who have at least a sixth-grade reading level),
* Diagnosed with psychiatric and neurological diseases,
* Diagnosed with dementia,
* Received chemotherapy treatment more than once,
* Planned to receive radiotherapy treatment together with chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline Anxiety level | baseline, 60-120 minute
  Baseline and post-intervention anxiety level assessed by trained research nurse using Spielberg's State-Trait Anxiety Inventory (STAI). The test scores between 20 and 80, with higher scores indicating more generalized and stronger anxiety.

SECONDARY OUTCOMES:
Nausea level | baseline, 60-120 minute
  Baseline and post-intervention nausea level assessed by trained research nurse using VAS (0 to 10; 0 means no nausea,10 means severe nausea).
Satisfaction level | 60-120 minute
  Post-intervention satisfaction level assessed by trained research nurse using VAS (0 to 10; 0 means not satisfied, 10 means very satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Uludag University Faculty of Medicine Hospital, The Outpatient Chemotherapy Unit, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dalli OE, Dogan DA, Pehlivan S, Yildirim Y, Evrensel T. The effect of two different types of music played to cancer patients during chemotherapy on anxiety, nausea, and satisfaction levels. Support Care Cancer. 2023 Nov 20;31(12):710. doi: 10.1007/s00520-023-08165-9. PMID 37982892